CLINICAL TRIAL: NCT02188030
Title: Individual Exercise Program for Industrial Workers With Complaints of the Arm, Neck, or Shoulder (CANS): Study Protocol for a Randomized Controlled Trial.
Brief Title: Individual and Group Exercise Program for Industrial Workers With CANS: Randomized Controlled Trial
Acronym: Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rosimeire Simprini Padula (Other)
Responsible Party: Sponsor-Investigator, Rosimeire Simprini Padula, PhD, Universidade Cidade de Sao Paulo
Organization: Universidade Cidade de Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 480.968
Record Dates: First submitted 2014-06-19; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Musculoskeletal Disorder of the Neck
Keywords: musculoskeletal symptom; industrial workers; physical-activity program; resistance training; randomized controlled trial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Exercise Training (GET). (Active Comparator): Group Exercise Program. The participants allocated into the GET Group will receive a general exercise training realized in group of workers. Each training session started with a five minute swarm-up by slowly moving the neck, upper back, shoulder, arms and hands through pain-free range of motion; followed by 30 minutes of stretching and strengthening exercises for neck, upper back, shoulder, arms and hands, performed in the standing posture, sitting or lying. For resistance exercise, will be adopted 3 sets of 10 repetitions with a load of 80% of 1 repetitions maximum 12. Dumbbells and elastic bands and will be used as accessories to perform the resistance exercises.
  Interventions: Other: Group Exercise Program
- Individual Exercise Training (Active Comparator): Individual Exercise Program. The participants allocated into the IET Group will receive a individual and specific strength training with seven different exercises, based in training programme describe by Andersen et al. and Sundstrup et al . During the intervention period, the training intensity were progressively increased according to the principle of periodization and progressive overload. Dumbbells and elastic bands and will be used as accessories to perform the resistance exercises. Experienced instructors supervised every other training session.
  Interventions: Other: Individual Exercise Program

INTERVENTIONS:
Other: Group Exercise Program — The participants allocated into the GET Group will receive a general exercise training realized in group of workers. Each training session started with a five minute swarm-up by slowly moving the neck, upper back, shoulder, arms and hands through pain-free range of motion; followed by 30 minutes of stretching and strengthening exercises for neck, upper back, shoulder, arms and hands, performed in the standing posture, sitting or lying. For resistance exercise, will be adopted 3 sets of 10 repetitions with a load of 80% of 1 repetitions maximum. Dumbbells and elastic bands and will be used as accessories to perform the resistance exercises.
  Arms: Group Exercise Training (GET).
Other: Individual Exercise Program — The participants allocated into the IET Group will receive a individual and specific strength training with seven different exercises, based in training programme describe by Andersen et al.3 and Sundstrup et al4.
  During the intervention period, the training intensity were progressively increased according to the principle of periodization and progressive overload5. Dumbbells and elastic bands and will be used as accessories to perform the resistance exercises. Experienced instructors supervised every other training session.
  Arms: Individual Exercise Training

SUMMARY:
This study is double-blinded RCT, whose aim is to assess if an individual exercise program is more effective to reduce complaints in neck, shoulders and arms that an group exercise program, in industrial workers.

The participants will be randomly allocated to receive 12 treatment sessions of individual exercise training (IET) or in group exercise training (GET). Sessions will last 30 minutes and will be held twice a week for 12 weeks. Participants will also be encouraged to continue the use of medicines and other health care.

DETAILED DESCRIPTION:
This study is double-blinded RCT. Participants will be recruited from employees of the companies and industries located in the South of Bahia, Brazil or by referral from general practitioners, orthopedists, This study is single-blinded RCT, whose aim is to assess the efficacy of an individual exercise program for employees with complaints in neck, shoulders and arms. Participants will be recruited from employees of the companies and industries located in Brazil or by referral from general practitioners, orthopedists, neurologists or physiatrists.

The sample of 100 participants was determined by a sample size calculation designed to detect a clinically important difference of 10 points in the DASH Questionnaire (estimated standard deviation = 16,65 points). The following specifications will be considered: α=0.05, statistical power of 80% and follow-up loss of up to 15%.

The participants will be randomly allocated to receive 12 treatment sessions of individual exercise training (IET) or in group exercise training (GET). Sessions will last 30 minutes and will be held twice a week for 12 weeks. Participants will also be encouraged to continue the use of medicines and other health care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnose of nontraumatic complaints of the arm, neck or shoulder with minimum intensity of 4 points on the visual analogue pain scale1, for at least 6 weeks2.

Exclusion Criteria:

* Participants with contraindication to physical exercise
* Participants who had been diagnosed with cervical disc hernia; shoulder instability; fractures; frozen shoulder; systemic diseases such as rheumatoid arthritis or diabetes; neurological diseases or other severe medical or psychiatric disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity during and after treatment | 6th and 12th week after the start of treatment
  Numeric Pain Rating Scale (NPRS) assesses the pain intensity levels perceived by the patient using likert 11-point scale (ranging from 0 to 10), with 0 representing "no pain" and 10 representing "the worst possible pain". The participants will be instructed to report the level of pain intensity in the last seven days.

SECONDARY OUTCOMES:
Global Impression of Recovery | 6th and 12th week after treatment
  The Global Perceived Effect Scale assesses the patient's perception, on a numerical scale, about how much their condition has improved or deteriorated comparing the onset of symptoms to the last few days. It is an 11-point numerical scale ranging -5 to +5, where the negative scores means that the patients are worsening, and the positive scores means refer positive that patients are recovering compared to the beginning. This scale has adequate clinimetric properties and it has been recommended for use as outcome measure for chronic pain trials 15.
Disability | Baseline, 6th and 12th week after treatment
  Disability Arm, Shoulder and Hand Questionnaire (DASH) is a questionnaire used to measure of disability and symptoms in the previous week of arm, shoulder and hand. The questionnaire uses a likert 5-point scale Likert (ranging from 1 to 5), with 1 means "no difficulty to perform, no symptom or no impact") and 5 means "unable to do, very severe symptom, or high impact". The total score ranges from 0 to 10, where 0 "no dysfunction" and 100 "severe impairment".

CONTACTS AND LOCATIONS:
Overall Officials: Rosimeire Padula, Doctor, Principal Investigator — Universidade Cidade de São Paulo (UNICID)
Locations (1):
- União Metropolitana de Ensino e Cultura (UNIME), Itabuna, Estado de Bahia, Brazil